CLINICAL TRIAL: NCT06595303
Title: Feelings of Patients Who Received Nitrous Oxide During Childbirth
Brief Title: Nitrous Oxyde During Labour
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SRB2024218
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Nitrous Oxide; Labour Analgesia
Keywords: Nitrous oxide; labour analgesia
MeSH Terms: interventions — Nitrous Oxide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- N2O for labour analgesia: Any woman who received nitrous oxide for childbirth at Hôpital Érasme between October 1, 2024 and April 30, 2025 and who signed the informed consent form for this study.
  Interventions: Drug: Nitrous oxide for labour analgesia

INTERVENTIONS:
Drug: Nitrous oxide for labour analgesia — Any woman may choose to have nitrous oxide inhalation as a standard protocol for labour analgesia

SUMMARY:
1. Background to the clinical research project Nitrous oxide is a valuable tool in medicine for its rapid and effective analgesic and sedative properties. It is used in 50% gaseous form for painful procedures. One frequent application is obstetric analgesia. However, in addition to its analgesic effects, many articles mention the psychotropic, even psychedelic, effects of nitrous oxide use. In one of the most recent studies, entitled More than just joy: A qualitative analysis of participant experiences during nitrous oxide sedation, involving healthy volunteers, it is reported that the sensations and feelings of the subjects are not necessarily pleasant, and many volunteers report psychedelic-like sensations, dreams or disturbed perceptions. The authors then question whether these effects are due to an absence of painful stimuli and therefore an absence of a beneficial effect. The same effects have been reported by Atkinson et al, also on volunteer subjects. Parturients feelings are highly variable, with a stronger focus on analgesic efficacy.
2. Objectives of the clinical research project 2.1 Primary objective: The main objective will be to evaluate the effects of nitrous oxide, other than analgesia, in the specific context of childbirth. The study will focus mainly on subjective feelings, as well as the effects of disconnection from reality.

   2.2 Secondary objectives: As secondary objectives, we will study the efficacy on pain.
3. Methodology of the clinical research project All patients who have received nitrous oxide for delivery as part of the standard course of treatment in the delivery room will be contacted within 24 hours by one of the investigators. The protocol, i.e. the questionnaire, will be explained to the patients and, if they accept the protocol, written consent will be obtained. Patients will then complete the questionnaire in the presence of one of the investigators, who will be able to explain the questions if necessary. The questionnaire will take around 20 minutes to complete.
4. Design of the clinical research project Prospective study based on a questionnaire.
5. Participants Any person who received nitrous oxide for childbirth at Hôpital Érasme between October 1, 2024 and April 30, 2025 and who signed the informed consent form for this study.

ELIGIBILITY:
Inclusion Criteria:

* Any person who received nitrous oxide for childbirth at Hôpital Érasme between October 1, 2024 and April 30, 2025 and who signed the informed consent form for this study.

Exclusion Criteria:

* No informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women in labour
Study Population: Any woman who received nitrous oxide for childbirth at Hôpital Érasme between October 1, 2024 and April 30, 2025 and who signed the consent form for this study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Unpleasant psychotropic effects | 12 hours
  Percentage (%) of patients who report an unpleasant psychotropic effect during nitrous oxide administration for labour analgesia.

SECONDARY OUTCOMES:
Analgesic effect | 12 hours
  All patients will report the analgesic efficiency of nitrous oxide during labour analgesia using a 3 point scale (very effective - somewhat effective - no effect). Percentage (%) of each effect will be presented.

CONTACTS AND LOCATIONS:
Locations (1):
- H.U.B - Hôpital Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carles G. [Pregnancy, delivery and customs: transcultural approach in obstetrics]. J Gynecol Obstet Biol Reprod (Paris). 2014 Apr;43(4):275-80. doi: 10.1016/j.jgyn.2013.12.002. Epub 2014 Jan 17. French. PMID 24440128
- [Background] Waldenstrom U, Hildingsson I, Rubertsson C, Radestad I. A negative birth experience: prevalence and risk factors in a national sample. Birth. 2004 Mar;31(1):17-27. doi: 10.1111/j.0730-7659.2004.0270.x. PMID 15015989
- [Background] Richardson MG, Raymond BL, Baysinger CL, Kook BT, Chestnut DH. A qualitative analysis of parturients' experiences using nitrous oxide for labor analgesia: It is not just about pain relief. Birth. 2019 Mar;46(1):97-104. doi: 10.1111/birt.12374. Epub 2018 Jul 22. PMID 30033596
- [Background] Valtonen P, Markkanen S, Jarventausta K, Tenhunen M, Kalliomaki ML. More than just joy: A qualitative analysis of participant experiences during nitrous oxide sedation. Acta Anaesthesiol Scand. 2024 Aug;68(7):906-912. doi: 10.1111/aas.14428. Epub 2024 Apr 9. PMID 38594960
- [Background] Atkinson RM, Green JD, Chenoweth DE, Atkinson JH. Subjective effects of nitrous oxide: cognitive, emotional, perceptual and transcendental experiences. J Psychedelic Drugs. 1979 Oct-Dec;11(4):317-30. doi: 10.1080/02791072.1979.10471415. No abstract available. PMID 522172
- [Background] Block RI, Ghoneim MM, Kumar V, Pathak D. Psychedelic effects of a subanesthetic concentration of nitrous oxide. Anesth Prog. 1990 Nov-Dec;37(6):271-6. PMID 2097905
- [Background] Migliaccio L, Lawton R, Leeman L, Holbrook A. Initiating Intrapartum Nitrous Oxide in an Academic Hospital: Considerations and Challenges. J Midwifery Womens Health. 2017 May;62(3):358-362. doi: 10.1111/jmwh.12635. Epub 2017 May 29. PMID 28556573
- [Background] Moon JS, Kuza CM, Desai MS. William James, Nitrous Oxide, and the Anaesthetic Revelation. J Anesth Hist. 2018 Jan;4(1):1-6. doi: 10.1016/j.janh.2017.10.012. Epub 2017 Dec 1. PMID 29559088
- [Background] Kronenberg G, Seifritz E, Olbrich S. Nitrous oxide inhalation: History and experiences. Acta Anaesthesiol Scand. 2024 Sep;68(8):1129. doi: 10.1111/aas.14462. Epub 2024 May 30. No abstract available. PMID 38815989
- [Background] Husum B, Stenqvist O, Alahuhta S, Sigurdsson GH, Dale O. Current use of nitrous oxide in public hospitals in Scandinavian countries. Acta Anaesthesiol Scand. 2013 Oct;57(9):1131-7. doi: 10.1111/aas.12165. Epub 2013 Jul 29. PMID 23889322